CLINICAL TRIAL: NCT02202642
Title: The Improvement of Limbal Epithelial Culture Technique for the Treatment of Unilateral Limbal Insufficiency by Using Collagenase to Isolate Limbal Stem Cells
Brief Title: The Improvement of Limbal Epithelial Culture Technique by Using Collagenase to Isolate Limbal Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Wei-Li Chen/Assistant Professor, National Taiwan University, Department of Ophthalmology., National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201007032D
Record Dates: First submitted 2011-04-21; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Alkaline Chemical Burn Of Cornea And Conjunctival Sac; Acid Chemical Burn Of Cornea And Conjunctival Sac; Benign Mucous Membrane Pemphigoid With Ocular Involvement
MeSH Terms: interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- limbal stem cells (Experimental): Using collagenase to isolate limbal stem cells and improve the technique of ex vivo expansion of limbal stem cells for the treatment of patients suffering from unilateral limbal stem cell insufficiency based on the concept of "limbal stem cells need special cell-cell contact and cell-extracellular matrix interaction to support their survival"
  Interventions: Procedure: collagenase

INTERVENTIONS:
Procedure: collagenase — Cultured limbal stem cells transplantation

SUMMARY:
Using collagenase to isolate limbal stem cells and improve the technique of ex vivo expansion of limbal stem cells for the treatment of patients suffering from unilateral limbal stem cell insufficiency based on the concept of "limbal stem cells need special cell-cell contact and cell-extracellular matrix interaction to support their survival".

DETAILED DESCRIPTION:
Patients suffering from unilateral limbal stem cell insufficiency and understand the benefits and risk factors of the operation will be enrolled in this clinical trial. Two weeks before transplantation, the investigators first take 1-2 mm2 of limbal tissues from the healthy eye, digest the tissue with collagenase, and get an epithelial cell cluster. The cell cluster will be cultured on amniotic membrane with SHEM medium which contains Dulbecco's modified Eagle's medium/F12 (1:1), 5% dimethyl sulfoxide, 10 ng/ml human epidermal growth factor, 5μg/ml insulin, 0.5 μg/ml hydrocortisone, 1 nM cholera toxin, 50μg/ml gentamicin, 1.25μg/ml amphotericin B. Seven to ten days later after successful culture, transplantation will be performed after the cells reaches 1.5-2 cm2 compact confluent epithelial sheets without evidence of contamination. During the operation, lamellar keratectomy will be performed to remove the abnormal corneal neovascularization and scar tissue. The cultivated epithelial sheets will be transplanted to denuded corneal surface with fibrin glue and suture technique. The patients are planed to be admitted for 2 weeks. After discharge, follow up of the patients will be performed on one week, two week, one month, two months, three months, six months and one year later. Pictures of external eyes will be taken and the extent of corneal epithelium regeneration, visual acuity, and complications will be recorded during follow-up visits. The investigators plan to collect 10 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 18-70 years old.
2. Lesion eye should have limbal insufficiency more than 180 degrees.
3. Lesion eye should have recurrent corneal erosions, corneal neovascularisation and poor vision caused by limbal insufficiency.
4. The symptoms should be more than 1/2 year, and have no possibility of improvement by medical treatment.
5. The patients will to received the operation and the long term post- operative follow-up.
6. The patients are not infected by AIDS, hepatitis B/C , and willing to received the associated examinations.
7. The patients does not plan to be pregnant from the day of cell culture and transplantation for 1 year. They also agree to receive the pregnant test.
8. The condition of cell culture from the 1st to the clinical trial is successful.

Exclusion Criteria:

1. Bilateral limbal insufficiency.
2. No recurrent corneal erosion, corneal neovascularisation or poor vision was found due to limbal insufficiency. If corneal neovascularisation was found deeper than the anterior 1/2 of corneal stroma, or corneal thickness was less than 200 um evaluated by anterior segment OCT and ultrasound pachymetry, the patients should be excluded from the operation criteria. If corneal thickness becomes thicker, the patients can be enrolled for operation.
3. About corneal sedation, if the value checked by Cocet-Bonnet esthesiometer is less than 5 mm, the patients should be excluded from operation.
4. The condition can be improved by medication, or resolve spontaneously.
5. Post-operative follow up is less than 1/2 year
6. The patient can't receive long term postoperative follow up
7. No light perception, or can be expected to have very poor prognosis
8. If the intraocular pressure was more than 21 mmHg under necessary glaucoma surgery and anti-glaucoma medication, or optic disc cupping was more than 90%, or visual field was found to have severe defects, the patients were excluded from the clinical trial.
9. Severe lagophthalmos or trichiasis, and does not received blepharoplasty.
10. Severe dry eye syndrome. Those patients with schirmer's test result less than 1 mm should be excluded.
11. If the cells in the first part of the clinical trial can't be successfully cultivated, the patients should be excluded. If the patients insisted to received further treatment, they can be enrolled 3 months later.
12. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Using collagenase to isolate limbal stem cells and improve the technique of ex vivo expansion of limbal stem cells for the treatment. | 12 months
  Nine to twelve days later after successful culture, transplantation will be performed after the cells diameter reaches 1.5-2.0 cm compact confluent epithelial sheets without evidence of contamination.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Li Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wei-Li Chen, Taipei, Taiwan